CLINICAL TRIAL: NCT00639912
Title: Randomized Trial on the Effects of Hydration With Sodium Chloride Versus Sodium Bicarbonate to Prevent Contrast Induced Nephropathy, in Patients Undergoing Primary Coronary Interventions for Acute ST Elevation Myocardial Infarction.
Brief Title: Effects of Hydration to Prevent Contrast Induced Nephropathy in PCI for ST-elevation Myocardial Infarction.
Acronym: CINIMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: Azienda Sanitaria Ospedaliera (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAN1374
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2025-06-11 (Actual); Status verified 2008-03

CONDITIONS: Contrast Induced Nephropathy
Keywords: contrast induced nephropathy STEMI PCI
MeSH Terms: interventions — Sodium Chloride; Sodium Bicarbonate; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A: low volume saline (Active Comparator): Solution of 154 mEq/L of sodium chloride. Rate of infusion: 1 ml/kg/hour for 12 hours after the procedure, starting in the Cath Lab.
  Interventions: Drug: sodium chloride
- B: high volume saline (Active Comparator): Solution of 154 mEq/L of sodium chloride. Rate of infusion: 3 ml/Kg for 1 hour, followed by 1 ml/Kg/hour for 12 hours after the procedure, starting in the Cath lab.
  Interventions: Drug: sodium chloride
- C: low volume sodium bicarbonate (Active Comparator): Solution of 154 mEq/L of sodium bicarbonate. Rate of infusion: 1 ml/Kg/hour for 12 hours after the procedure, starting in the Cath Lab.
  Interventions: Drug: sodium bicarbonate
- D: high volume sodium bicarbonate (Active Comparator): Solution of 154 mEq/L of sodium bicarbonate. Rate of infusion: 3 ml/Kg for 1 hour, followed by 1 ml/Kg/hour for 12 hours after the procedure, starting in the Cath Lab.
  Interventions: Drug: sodium bicarbonate

INTERVENTIONS:
Drug: sodium chloride — Solution of 154 mEq/L of sodium chloride. Rate of infusion: 1 ml/Kg/hour for 12 hours.
  Other Names: Normal saline. Isotonic saline. Sodium chloride 0.9% .
  Arms: A: low volume saline
Drug: sodium chloride — Solution of 154 mEq/L of sodium chloride. Rate of infusion: 3 ml/Kg for 1 hour, followed by 1 ml/Kg/hour for 12 hours
  Other Names: Normal saline. Isotonic saline. Sodium Chloride 0.9% .
  Arms: B: high volume saline
Drug: sodium bicarbonate — 154 mEq/L of sodium bicarbonate in dextrose solution. Rate of infusion: 1 ml/Kg/hour for 12 hours.
  Other Names: Addition of 77 ml 8,4% Na bicarbonate to 423 ml 5% dextrose.
  Arms: C: low volume sodium bicarbonate
Drug: sodium bicarbonate — 154 mEq/L of sodium chloride in dextrose solution. Rate of infusion: 3 ml/Kg for 1 hour, followed by 1 ml/Kg/hour for 12 hours.
  Other Names: Addition of 77 ml 8,4% Na bicarbonate to 423 ml 5% dextrose.
  Arms: D: high volume sodium bicarbonate

SUMMARY:
The aim of the study is to test the efficacy of low versus high volume hydration and two different solutions (sodium chloride versus sodium bicarbonate) in preventing contrast induced nephropathy (CIN) in ST elevation myocardial infarction (STEMI) patients undergoing primary PCI.

DETAILED DESCRIPTION:
Contrast-induced nephropathy (CIN) is associated with increased morbidity and mortality after percutaneous coronary interventions (PCI). Patients with ST elevation myocardial infarction (STEMI) are at high risk for CIN because of hemodynamic instability of the patient, inability to prevent the phenomenon (hydration) and the possible exposure to high volume of contrast media. Recent reports have shown incidence of CIN up to 19% in this population and a related increase of in-hospital mortality.

Merten e coll. (JAMA 2004) reported that sodium bicarbonate infusion before and after contrast exposure in patients with chronic renal failure and without myocardial infarction (AMI) is more effective than sodium chloride in preventing CIN.

Up to date there is no evidence of any effective prophylactic measures in patients with STEMI undergoing primary PCI.

The aim of the study is to test the efficacy of low versus high volume hydration and the efficacy of two different solutions (sodium chloride versus sodium bicarbonate) in preventing CIN in STEMI patients undergoing primary PCI.

The infusion of the randomized solution will start just after randomization and after determination of baseline serum creatinine.

Determination of serum creatinine will be repeated at 24, 48 and 72 hours after randomization. Creatinine clearance will be calculated with Cockroft-Gault formula and MDRD.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of years
* Chest pain lasting at least 30 minutes, non responsive to nitrates, associated to ST elevation of at least 0.2 mV on surface ECG in two or more contiguous leads or to new left bundle branch block.
* Informed consent

Exclusion Criteria:

* Chronic hemodialytic or peritoneal treatment
* Coronary anatomy unsuitable for PCI
* Need of emergency coronary artery by-pass grafting
* Post-anoxic coma
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2007-06; Primary Completion 2010-05 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
contrast induced nephropathy incidence | 24, 48 and 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Manari, MD, Principal Investigator — Arcispedale S. Maria Nuova Reggio Emilia
Locations (5):
- Italy (5):
  - Azienda Ospedaliera Universitaria S. Anna, Ferrara, Emilia-Romagna
  - Nuovo Ospedale Civile di Baggiovara, Modena, Emilia-Romagna
  - Arcispedale S. Maria Nuova, Reggio Emilia, Emilia-Romagna
  - Dipartimento di Cardiologia, Ospedale di Lavagna, Lavagna, Genova
  - Dipartimento di Cardiologia, Ospedale Maggiore, Parma, Parma

REFERENCES:
- [Background] McCullough PA, Adam A, Becker CR, Davidson C, Lameire N, Stacul F, Tumlin J; CIN Consensus Working Panel. Risk prediction of contrast-induced nephropathy. Am J Cardiol. 2006 Sep 18;98(6A):27K-36K. doi: 10.1016/j.amjcard.2006.01.022. Epub 2006 Feb 23. PMID 16949378
- [Background] Marenzi G, Lauri G, Assanelli E, Campodonico J, De Metrio M, Marana I, Grazi M, Veglia F, Bartorelli AL. Contrast-induced nephropathy in patients undergoing primary angioplasty for acute myocardial infarction. J Am Coll Cardiol. 2004 Nov 2;44(9):1780-5. doi: 10.1016/j.jacc.2004.07.043. PMID 15519007
- [Background] Marenzi G, Assanelli E, Marana I, Lauri G, Campodonico J, Grazi M, De Metrio M, Galli S, Fabbiocchi F, Montorsi P, Veglia F, Bartorelli AL. N-acetylcysteine and contrast-induced nephropathy in primary angioplasty. N Engl J Med. 2006 Jun 29;354(26):2773-82. doi: 10.1056/NEJMoa054209. PMID 16807414
- [Background] Merten GJ, Burgess WP, Gray LV, Holleman JH, Roush TS, Kowalchuk GJ, Bersin RM, Van Moore A, Simonton CA 3rd, Rittase RA, Norton HJ, Kennedy TP. Prevention of contrast-induced nephropathy with sodium bicarbonate: a randomized controlled trial. JAMA. 2004 May 19;291(19):2328-34. doi: 10.1001/jama.291.19.2328. PMID 15150204
- [Derived] Manari A, Magnavacchi P, Puggioni E, Vignali L, Fiaccadori E, Menozzi M, Tondi S, Robotti S, Ferrari D, Valgimigli M. Acute kidney injury after primary angioplasty: effect of different hydration treatments. J Cardiovasc Med (Hagerstown). 2014 Jan;15(1):60-7. doi: 10.2459/JCM.0b013e3283641bb8. PMID 24500238